CLINICAL TRIAL: NCT06329271
Title: Compare Early Weight Bearing as Tolerated (WBAT) Group With Weight Bearing Restriction(WBR) After Hip Fracture Nailing,
Brief Title: After Hip Fracture Nailing, Compare Early Weight Bearing as Tolerated (WBAT) Group With Weight Bearing Restriction(WBR)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 113022-E
Record Dates: First submitted 2024-03-18; First posted 2024-03-25 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2024-03

CONDITIONS: Bony Weight Bearing Disorder
Keywords: fracture reduction; proximal femur fracture; geriatrics; early weight-bearing
MeSH Terms: conditions — Proximal Femoral Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early-Weight bearing (Experimental): Early Weight bearing was defined as starting Weight bearing within 48 h postoperatively, and WBAT referred to the adjustment of fracture site weight-bearing by pain tolerance.
  Interventions: Behavioral: Early-Weight bearing
- Weight-bearing restriction (No Intervention): Weight bearing as toleration started after 48 h postoperatively.

INTERVENTIONS:
Behavioral: Early-Weight bearing — The patients began early weight bearing under attending physician and physiotherapist surveillance within 48 hours after surgery. Patients were instructed to stand up near the bed, and muscle power, gait stability, and pain tolerance were recorded. The physiotherapist instructed the patients to perform early mobilization and weight bearing as tolerable by self-adjustment of body weight distribution over the bilateral lower extremities, and walking assistance was used to prevent repeat falling accidents.
  Arms: Early-Weight bearing

SUMMARY:
Purpose: Proximal femur fracture is a major traumatic injury in elderly populations; however, practical postoperative weight-bearing protocols are lacking. Therefore, the purpose of the present study was to investigate whether early weight-bearing status after proximal femur nail fixation is associated with any loss of reduction and evaluate the clinical outcomes of this intervention.

Patients and methods:

For this prospective single-center clinical trial study, we recruited 60 geriatric proximal femur fracture cases, classified by AO/OTA 2018, receiving intramedullary nail fixation. The participants were assigned to the Early-weight-bearing group (n= 30) or the Weight-bearing restriction group (n = 30). Clinical outcomes included the Harris functional hip score and VAS pain score. Additionally, demographic data, radiological parameters, time to weight-bearing, mortality rate, medical and surgical complications, and final ambulation status were recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patients with AO/OTA type 31 fractures were included, and all fractures were classified using intraoperative fluoroscopy with traction on the fracture table.

Exclusion Criteria:

* Patients with pathological fractures, neurovascular insufficiency, ipsilateral lower extremity musculoskeletal injury, multiple fractures, or high risk of falling, including frequent falling accidents within 6 months, unsteady gait, ipsilateral neuropathy, limb weakness, and urinary incontinence were excluded.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-03-08 (Actual); Primary Completion 2025-04-29 (Estimated); Study Completion 2025-04-29 (Estimated)

PRIMARY OUTCOMES:
Harris Hip Functional score | Functional and radiographic evaluations was performed at week 1 postoperatively
  The questionaire to patient. (HHS score 0-100,<60 poor,>80 good)
Harris Hip Functional score | Functional and radiographic evaluations was performed at months 1 postoperatively
  The questionaire to patient. (HHS score 0-100,<60 poor,>80 good)
Harris Hip Functional score | Functional and radiographic evaluations was performed at months 3 postoperatively
  The questionaire to patient. (HHS score 0-100,<60 poor,>80 good)
Harris Hip Functional score | Functional and radiographic evaluations was performed at months 6 postoperatively
  The questionaire to patient. (HHS score 0-100,<60 poor,>80 good)
Harris Hip Functional score | Functional and radiographic evaluations was performed at months 12 postoperatively
  The questionaire to patient. (HHS score 0-100,<60 poor,>80 good)

SECONDARY OUTCOMES:
Visual analog pain score | Record at week 1 postoperatively
  Independent assessor (VAS:0-10, higher scores mean a worse outcome)
Visual analog pain score | Record at months 1 postoperatively
  Independent assessor (VAS:0-10, higher scores mean a worse outcome)
Visual analog pain score | Record at months 3 postoperatively
  Independent assessor (VAS:0-10, higher scores mean a worse outcome)
Visual analog pain score | Record at months 6 postoperatively
  Independent assessor (VAS:0-10, higher scores mean a worse outcome)
Visual analog pain score | Record at months 12 postoperatively
  Independent assessor (VAS:0-10, higher scores mean a worse outcome)
Complication | Functional and radiographic evaluations were performed at week 1, months 1, 3, 6, and 12 postoperatively
  Loss of reduction, malunion, nonunion or medical complications

CONTACTS AND LOCATIONS:
Locations (1):
- Far-Eastern Memorial Hospital, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided